CLINICAL TRIAL: NCT06983574
Title: Evaluating the Effectiveness of an mHealth Application to Promote Home-Based Exercise in Adults Aged 65 and Older: A Randomized Controlled Trial
Brief Title: Effectiveness of an mHealth Application to Promote Home-Based Exercise in Adults Aged 65 and Older
Acronym: HOME-FIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PXL University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HOME-FIT
Record Dates: First submitted 2025-05-12; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIA intervention (Experimental): Participants will use the mHealth app to engage in home-based workouts aimed at promoting physical activity. The app provides exercises lasting approximately 12-15 minutes each, which participants are encouraged to perform regularly to achieve a total of at least 150 minutes of moderate-to-vigorous physical activity per week. The intervention period spans 8 weeks, during which participants should follow the app's guidance to complete the recommended workouts and track their progress. Participan
  Interventions: Other: MIA
- No intervention with MIA (No Intervention): Participants in the control group will be instructed to maintain their usual physical activity, dietary habits, and sleep patterns for the 8-week study duration. They will be asked to refrain from engaging in any specialized exercise training during this time.

INTERVENTIONS:
Other: MIA — Through a collaborative co-creation process, MIA, a mHealth app was developed and refined over multiple iterations with the goal of promoting physical activity and fostering a lifestyle centred around an active and healthy approach. Content and design were derived from both the co-creative workshops and based on the theoretical framework of the intervention functions of the BCW. The final mHealth app is composed by five major features:
  * Tailor-made tips
  * Literacy aiming to improve awareness about PA and an active healthy lifestyle
  * Exercise workouts
  * Community calendar aiming to enhance social connections
  * A diary consisting of daily activities (MIA workouts and self-registration) To customize the user experience, a brief personal description was created as the start screen, which prompts older adults to answer questions related to their baseline physical activity level, motivation, and medical history.
  Arms: MIA intervention

SUMMARY:
The goal of this clinical trial is to learn if drug ABC works to evaluate the effectiveness of an mHealth application to promote home-based exercise in adults aged 65 and older. The objectives are:

Primary objective:

• To evaluate the effect of the mHealth application on increasing moderate-to-vigorous physical activity levels.

Secondary objectives:

* To assess the impact of the mHealth application on physical fitness measures (e.g., functional capacity, strength, balance, fall risk, flexibility)
* To assess the impact of the mHealth application on physical activity (e.g., daily steps, self-reported physical activity)
* To examine the impact of the mHealth application on wellbeing
* To explore the impact of the mHealth application on cognitive functioning
* To measure user adherence and engagement with the mHealth application
* To evaluate participant satisfaction with the mHealth application

Researchers will compare a group using an mHealth application to a group not using the application to determine whether it effectively increases physical activity.

Participants will:

* Use the mHealth application or not for 8 weeks
* Visit the labo 3 times in total for assessements
* Use a wearable during the study period

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Medically stable Any existing chronic illnesses (e.g., hypertension, diabetes, or arthritis) are being effectively managed with medications or lifestyle interventions.

The participant is not experiencing any recent or ongoing acute medical conditions, such as infections, recent surgeries, or injuries, that could interfere with participation in the study.

* No significant cognitive, mental or physical impairment that would prevent safe use of the mHealth application or performance of the exercises.
* Understanding and speaking Dutch
* Access to a smartphone and computer.

Exclusion Criteria:

* The presence of an active lifestyle.
* Enrolment in other exercise programs or clinical trials that might interfere with study participation or outcomes.
* Any condition or circumstance deemed by a healthcare professional to pose a risk to the participant's safety or the validity of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
MVPA | From enrollment to 3 months post-intervention
  Moderate-to-vigorous physical activity (MVPA) will be assessed using a wearable activity tracker, the Garmin Vivomart 5, which allows for continuous, 24/7 monitoring of physical activity. This device tracks various types of movement throughout the day, providing comprehensive data on activity levels and enabling detailed analysis of participants' physical activity patterns over time.

SECONDARY OUTCOMES:
Gait speed | From enrollment to the end of intervention at 8 weeks
  Gait speed will be measured using the Six Minute Walking Test performed according to the ERS/ATS (22). The absolute distance walked in the test will be used for analysis, and compared with normative values.
Quadriceps force | From enrollment to the end of intervention at 8 weeks
  Isometric quadriceps force will be assessed using the Kinvent®2016 (Kinvent, Montpellier, France) handheld dynamometer. Participants will be tested while sitting in an upright position. The assessor applies resistance and askes the participant to maximally contract the muscle against the resistance. At least three maximal efforts will be performed and the test will be repeated until reproducible measurements (less than 10 % variability) are obtained. The highest value will be used for analyses and compared with normative values.
Handgrip strength | From enrollment to the end of intervention at 8 weeks
  Handgrip strength will be measured isometrically using the K-Force Grip® (Kinvent, Montpellier, France) while sitting in the upright position with the elbow flexed 90◦ and the wrist in a neutral position. Three maximal efforts will be performed and repeated until reproducible measurements (less than 10 % variability) will be obtained. The highest value will be used for analysis and compared with normative values.
Balance | From enrollment to the end of intervention at 8 weeks
  Postural balance will be assessed using the Kinvent PLATES v3® (Kinvent, Montpellier, France). Participants will undergo a double leg balance test three times for 10 seconds with eyes opened and eyes closed, followed by a single leg balance test consisting of three repetitions for each leg with eyes opened.
Fall risk | From enrollment to the end of intervention at 8 weeks
  The Timed Up & Go test will be conducted to evaluate fall risk. Participants will be observed and timed as they stand up from an armchair, walk three meters, turn around, walk back, and sit down again.
Flexibility | From enrollment to the end of intervention at 8 weeks
  The Sit and Reach test will assess the spinal flexibility and hamstring length/flexibility. Participants will be seated on the floor with their legs extended and feet placed flat against a sit-and-reach box. A measuring scale will be attached to the top of the box. With their hands placed on top of the other, participants will be instructed to reach forward toward their toes as far as possible. The distance reached will be recorded using the measuring scale. The highest value will be used for analysis.
Muscle power | From enrollment to the end of intervention at 8 weeks
  Muscle power will be assessed by the 30 s Sit-to-stand (STS) muscle power test. Briefly, the subjects will perform as many STS repetitions as possible in 30 s on a standardized armless chair from the sitting position-buttocks touching the chair-to the full standing position, with their arms crossed over the chest. Verbal encouragement will be given throughout the test. The participants will be allowed to try one to two times before the definitive measure was annotated.
Daily steps | From enrollment to 3 months post-intervention
  Daily steps will be assessed using a wearable activity tracker, the Garmin Vivomart 5.
IPAQ-SF | From enrollment to the end of intervention at 8 weeks
  The International Physical Activity Questionnaire - Short Form. The total score will be classified into three categories: low, moderate, and high physical activity, according to the IPAQ scoring guidelines.
ESES | From enrollment to the end of intervention at 8 weeks
  The Exercise Self-Efficacy Scale. The total score ranges between 10 and 40. Higher scores represent higher confidence to carry out physycial activity.
BREQ | From enrollment to the end of intervention at 8 weeks
  The Behavioural Regulations in Exercise Questionnaire. The total score will be transformed to a RAI score. Higher score represent higher self determination for physical activity.
PACES | From enrollment to the end of intervention at 8 weeks
  The Physical Activity Enjoyment Scale. The total score ranges between 8 and 56. Higher scores represent greater enjoyment for physical activity.
Cognitive function | From enrollment to the end of intervention at 8 weeks
  The assessment of cognitive functioning will be conducted using the SWAY (SWAY Medical Inc. in Tulsa, OK, USA). The cognitive performance segment of the app encompasses three modules focusing on memory, reaction time, and impulse control. Based on the results, participants will be classified into percentiles ranging from vary low (<10%) to very high (>10%).
WHO-QoL | From enrollment to the end of intervention at 8 weeks
  The World Health Organization Quality of Life questionnaire. The total score ranges between 0 and 100. Higher scores represent higher quality of life.
PSS | From enrollment to the end of intervention at 8 weeks
  The Perceived Stress Scale. The total score ranges between 0 and 40. Higher scores represent higher perceived stress.
GSQ | From enrollment to the end of intervention at 8 weeks
  The Geriatric Sleep Questionnaire. The total score ranges between 6 and 30. Higher scores represent poorer sleep quality.
SUS | From enrollment to the end of intervention at 8 weeks
  The System Usability Scale. The total score ranges between 1 and 100. Higher scores represent high usability.
NPS | From enrollment to the end of intervention at 8 weeks
  The Net Promoter Score. Total score ranges between 1 and 10. Higher scores represent higher loyalty.
CSAT | From enrollment to the end of intervention at 8 weeks
  The Customer Satisfaction Score. Total score ranges between 1 and 5. Higher scores represent higher satisfaction.

REFERENCES:
- [Derived] Quadflieg K, Robijns J, Daniels K. Evaluating the effectiveness of an mHealth application to promote home-based exercise in adults aged 65 years and older: protocol for a randomised controlled trial. BMJ Open. 2025 Nov 4;15(11):e106629. doi: 10.1136/bmjopen-2025-106629. PMID 41193218